CLINICAL TRIAL: NCT05212571
Title: Long-term Pain Modulation by Intravenous Esketamine in Complex Regional Pain Syndrome: a Non-inferiority Study
Brief Title: Long-term Pain Modulation by Intravenous Esketamine in CRPS
Acronym: KetCRPS-2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Thomas J. P. Mangnus, MD, Medical doctor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL77785.078.21; 2021-000640-21 (EudraCT Number); MEC-2021-0426 (Other: Medical Ethics Committee of Erasmus MC)
Record Dates: First submitted 2021-12-13; First posted 2022-01-28 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Complex Regional Pain Syndromes; CRPS (Complex Regional Pain Syndromes)
Keywords: CRPS; Complex Regional Pain Syndrome; ketamine; S-ketamine; esketamine
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Ketamine; Esketamine

STUDY DESIGN:
Intervention Model Description: prospective, randomized non-inferiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Outpatient (Experimental): The experimental intervention group visits the outpatient clinic to receive intravenous esketamine in day-care setting every 2 weeks for 3 months.
  Interventions: Drug: S-ketamine infusion outpatient setting
- Inpatient (Active Comparator): The standard treatment group receives intravenous esketamine for 6 consecutive days in hospital.
  Interventions: Drug: S-ketamine infusion inpatient setting

INTERVENTIONS:
Drug: S-ketamine infusion inpatient setting — S-ketamine is administered intravenously for six consecutive days. The administered dose of S-ketamine is 50 mcg/kg/h and can be increased to a maximum of 200 mcg/kg/h.
  Other Names: ketamine; esketamine
  Arms: Inpatient
Drug: S-ketamine infusion outpatient setting — S-ketamine is administered intravenously for six hours. The administered dose of S-ketamine is 50 mcg/kg/h and can be increased to a maximum of 200 mcg/kg/h.
  Other Names: ketamine; esketamine
  Arms: Outpatient

SUMMARY:
Intravenous administration of esketamine is an effective recognized therapeutic option in refractory pain in CRPS, which sometimes in at least a part of the patients has a prolonged therapeutic effect. Unfortunately, CRPS literature contains a wide range of ketamine dosing regimens with the result that clinical protocols on dosage and administration are very heterogeneous. The current esketamine regimen in Erasmus MC consists of a 6-day hospital admission for continuous administration. In the Netherlands, both inpatient and outpatient esketamine treatments are offered. Inpatient and outpatient ketamine treatments have never been compared in randomized controlled trials and it is therefore unknown whether these two dosing regimens are equally effective.

The primary objective is to demonstrate non-inferiority of experimental esketamine administration of 6x 1 day per 2 weeks (in total 3 months) as compared with standard esketamine administration of 1x 6 consecutive days. The end of study is at 6 months after the start of the study/treatment.

DETAILED DESCRIPTION:
Rationale: Complex regional pain syndrome (CRPS) is a debilitating chronic pain condition of one or more limbs. Its diagnosis is based on (combinations of) underlying pathophysiological mechanisms. Achieving relevant pain relief fails in a significant proportion of CRPS patients. Intravenous administration of esketamine is an effective therapeutic option in refractory pain in CRPS, which in at least a part of the patients has a prolonged therapeutic effect. Unfortunately, CRPS literature contains a wide range of ketamine dosing regimens with the result that clinical protocols on dosage and administration are very heterogeneous. In the Netherlands, both inpatient and outpatient esketamine treatments are offered. The current esketamine regimen in Erasmus MC consists of a 6-day hospital admission for continuous administration; however, logistical boundaries limit this therapy. Esketamine infusions in an outpatient setting might increase flexibility and availability of esketamine treatment. However, inpatient and outpatient ketamine treatments have never been compared in randomized controlled trials and it is therefore unknown whether these two dosing regimens are equally effective.

Objective: The primary objective is to demonstrate non-inferiority of experimental esketamine administration of 6x 1 day per 2 weeks (in total 3 months) as compared with standard esketamine administration of 1x 6 consecutive days at 3 months after the start of the study/treatment. The secondary objective is to assess pain scores till 6 months follow-up, logistical problems, adverse effects, questionnaires, thermography and quantitative sensory testing in both treatment groups.

Study design: Prospective, randomized, non-inferiority study in 60 patients

Study population: Sixty adult patients with chronic pain due to CRPS

Intervention: All patients will receive intravenous esketamine. The standard treatment group receives intravenous esketamine for 6 consecutive days (in hospital). The experimental intervention group visits the outpatient clinic to receive intravenous esketamine in day-care setting every 2 weeks for 3 months.

Main study parameters/endpoints: The main study parameter is pain intensity, measured by means of Numerical Rating Scale (NRS), to demonstrate non-inferiority of the experimental treatment after three months.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the new International Association for the Study of Pain (IASP) diagnostic criteria for CRPS ("the Budapest Criteria) (Harden et al., 2010) or having met the new IASP diagnostic criteria of CRPS ("CRPS with Remission of Some features") (Goebel et al., 2021).
* Willing and capable to participate in the study.
* CRPS in one upper extremity and/or CRPS in one lower extremity
* Treatment in an elective setting.
* Adequate comprehension of the Dutch language
* Age ≥ 18 years

Exclusion Criteria:

* Severe liver disease
* Psychiatric (schizophrenia, psychosis, delirium, manic depression)
* Active substance abuse
* Intoxication with alcohol or other substances
* Poorly controlled hypertension
* Unstable angina
* High-risk coronary vascular disease
* Heart failure
* Elevated intracranial pressure
* Elevated intraocular pressure
* Thyrotoxicosis
* Pregnancy
* Combination with derivates of xanthines (theophylline) or ergometrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain scores | Baseline (week 0), During inpatient or outpatient esketamine infusion (week 1 for inpatient protocol / week 1, 3, 5, 7, 9, 11 for outpatient protocol), During telephone consultation (week 1, 3, 5, 7, 9, 11), Follow-up (3 months), End of study (6 months)
  Pain intensity measured by Numerical Rating Scale (NRS). Minimum value=0 and maximum value is 10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from baseline Quantitative Sensory Testing | Baseline (week 0) and follow-up visit (week 12)
  To assess the sensory-discriminative dimensions of pain before and after ketamine treatment
Change from baseline Thermography | Baseline (week 0) and follow-up visit (week 12)
  Objectively measured effects on the extremity temperature by each of the administration regimens on symptoms vasomotor disturbances. The investigators use an infrared camera.
Adverse events due to S-ketamine infusion | During inpatient or outpatient esketamine infusion (week 1 for inpatient protocol / week 1, 3, 5, 7, 9, 11 for outpatient protocol), During telephone consultation (week 1, 3, 5, 7, 9, 11)
  Assessed by physical examination and vital parameters (blood pressure, heart rate, saturation and temperature)
Change from baseline pain medication dose | Baseline (week 0), follow-up visit (3 months) and end of study (6 months)
Change from baseline Complex Regional Pain Syndrome severity score | Baseline (week 0) and follow-up visit (3 months)
  according to Harden et al. (2010). All symptoms and signs are scored as Yes = 1 and No = 0. Sum up the total score (i.e., number of "Yes" responses) to derive the total CSS score. The Complex Severity Score can range from 0-16. Higher scores mean a worse outcome.
Global Perceived Effect | During telephone consultation (week 1, 3, 5, 7, 9, 11), follow-up visit (3 months) and end of study (6 months)
  The Global Perceived Effect asks the patient to rate, on a numerical scale 0-7, how much their condition has improved or deteriorated since some predefined time point. Higher scores mean a worse outcome. According to Hudak et al. 2000.
Patient-Reported Outcomes Measurement Information System (PROMIS) -29 Profile | Baseline (week 0) and follow-up visit (3 months)
  Assesses 7 domains, each with 4 questions (ranging from 1-5, ranging from no/never/not at all to yes/always/continuously): depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. According to Terwee et al. 2014
Short-form McGill Pain Questionnaire-2 | Baseline (week 0) and follow-up visit (3 months)
  Neuropathic pain items capturing the quality of pain. Scale ranging from 0-10. Higher scores mean a worse outcome. According to Dworkin et al., 2009
Pain Catastrophizing Scale | Baseline (week 0) and follow-up visit (3 months)
  The respondent considers how confident they are performing each activity, while taking their pain into account. Scale from 0-4. Higher scores mean a worse outcome. According to Sullivan et al., 2011
EQ-5D-5L. | Baseline (week 0) and follow-up visit (3 months)
  To measure health state, comprising mobility, self-care, usual activities, pain/discomfort, anxiety/depression.
  The 5 questions about health status are scored on a 5-point scale (1-5) Placing these numbers one after the other creates a 5-digit index that represents a health profile (eg 12323). According to Herdman et al., 2011
Pain Self-Efficacy Questionnaire | Baseline (week 0) and follow-up visit (3 months)
  The respondent considers how confident they are performing each activity, while taking their pain into account. The scale ranges from 0-6. Higher scores mean a better outcome. According to Nicholas et al., 2007

CONTACTS AND LOCATIONS:
Overall Officials: Frank JP Huygen, MD, PhD, Principal Investigator — Erasmus MC, Center for Pain Medicine; Thomas Mangnus, MD, Study Director — Erasmus MC, Center for Pain Medicine
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sigtermans MJ, van Hilten JJ, Bauer MCR, Arbous SM, Marinus J, Sarton EY, Dahan A. Ketamine produces effective and long-term pain relief in patients with Complex Regional Pain Syndrome Type 1. Pain. 2009 Oct;145(3):304-311. doi: 10.1016/j.pain.2009.06.023. Epub 2009 Jul 14. PMID 19604642
- [Background] Mangnus TJP, Bharwani KD, Stronks DL, Dirckx M, Huygen FJPM. Ketamine therapy for chronic pain in The Netherlands: a nationwide survey. Scand J Pain. 2021 Aug 24;22(1):97-105. doi: 10.1515/sjpain-2021-0079. Print 2022 Jan 27. PMID 34432970
- [Background] Mangnus TJP, Dirckx M, Bharwani KD, de Vos CC, Frankema SPG, Stronks DL, Huygen FJPM. Effect of intravenous low-dose S-ketamine on pain in patients with Complex Regional Pain Syndrome: A retrospective cohort study. Pain Pract. 2021 Nov;21(8):890-897. doi: 10.1111/papr.13056. Epub 2021 Jul 24. PMID 34233070
- [Background] Harden NR, Bruehl S, Perez RSGM, Birklein F, Marinus J, Maihofner C, Lubenow T, Buvanendran A, Mackey S, Graciosa J, Mogilevski M, Ramsden C, Chont M, Vatine JJ. Validation of proposed diagnostic criteria (the "Budapest Criteria") for Complex Regional Pain Syndrome. Pain. 2010 Aug;150(2):268-274. doi: 10.1016/j.pain.2010.04.030. Epub 2010 May 20. PMID 20493633
- [Background] Grieve S, Perez RSGM, Birklein F, Brunner F, Bruehl S, Harden RN, Packham T, Gobeil F, Haigh R, Holly J, Terkelsen A, Davies L, Lewis J, Thomassen I, Connett R, Worth T, Vatine JJ, McCabe CS. Recommendations for a first Core Outcome Measurement set for complex regional PAin syndrome Clinical sTudies (COMPACT). Pain. 2017 Jun;158(6):1083-1090. doi: 10.1097/j.pain.0000000000000866. PMID 28178071
- [Background] Goebel A, Birklein F, Brunner F, Clark JD, Gierthmuhlen J, Harden N, Huygen F, Knudsen L, McCabe C, Lewis J, Maihofner C, Magerl W, Moseley GL, Terkelsen A, Thomassen I, Bruehl S. The Valencia consensus-based adaptation of the IASP complex regional pain syndrome diagnostic criteria. Pain. 2021 Sep 1;162(9):2346-2348. doi: 10.1097/j.pain.0000000000002245. No abstract available. PMID 33729210
- [Background] Cohen SP, Bhatia A, Buvanendran A, Schwenk ES, Wasan AD, Hurley RW, Viscusi ER, Narouze S, Davis FN, Ritchie EC, Lubenow TR, Hooten WM. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Chronic Pain From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):521-546. doi: 10.1097/AAP.0000000000000808. PMID 29870458
- [Background] Zhao J, Wang Y, Wang D. The Effect of Ketamine Infusion in the Treatment of Complex Regional Pain Syndrome: a Systemic Review and Meta-analysis. Curr Pain Headache Rep. 2018 Feb 5;22(2):12. doi: 10.1007/s11916-018-0664-x. PMID 29404715
- [Background] Harden NR, Bruehl S, Perez RSGM, Birklein F, Marinus J, Maihofner C, Lubenow T, Buvanendran A, Mackey S, Graciosa J, Mogilevski M, Ramsden C, Schlereth T, Chont M, Vatine JJ. Development of a severity score for CRPS. Pain. 2010 Dec;151(3):870-876. doi: 10.1016/j.pain.2010.09.031. Epub 2010 Oct 20. PMID 20965657
- [Background] Hudak PL, Wright JG. The characteristics of patient satisfaction measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3167-77. doi: 10.1097/00007632-200012150-00012. PMID 11124733
- [Background] Terwee CB, Roorda LD, de Vet HC, Dekker J, Westhovens R, van Leeuwen J, Cella D, Correia H, Arnold B, Perez B, Boers M. Dutch-Flemish translation of 17 item banks from the patient-reported outcomes measurement information system (PROMIS). Qual Life Res. 2014 Aug;23(6):1733-41. doi: 10.1007/s11136-013-0611-6. Epub 2014 Jan 9. PMID 24402179
- [Background] Dworkin RH, Turk DC, Revicki DA, Harding G, Coyne KS, Peirce-Sandner S, Bhagwat D, Everton D, Burke LB, Cowan P, Farrar JT, Hertz S, Max MB, Rappaport BA, Melzack R. Development and initial validation of an expanded and revised version of the Short-form McGill Pain Questionnaire (SF-MPQ-2). Pain. 2009 Jul;144(1-2):35-42. doi: 10.1016/j.pain.2009.02.007. Epub 2009 Apr 7. PMID 19356853
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Mangnus TJP, Bharwani KD, Dirckx M, Huygen FJPM. From a Symptom-Based to a Mechanism-Based Pharmacotherapeutic Treatment in Complex Regional Pain Syndrome. Drugs. 2022 Apr;82(5):511-531. doi: 10.1007/s40265-022-01685-4. Epub 2022 Mar 5. PMID 35247200
- [Result] Mangnus TJP, Dirckx M, Bharwani KD, Baart SJ, Siepman TAM, Redekop K, Dik WA, de Vos CC, Huygen FJPM. Intermittent versus continuous esketamine infusions for long-term pain modulation in complex regional pain syndrome: protocol of a randomized controlled non-inferiority study (KetCRPS-2). BMC Musculoskelet Disord. 2023 Mar 29;24(1):239. doi: 10.1186/s12891-023-06258-4. PMID 36991381